CLINICAL TRIAL: NCT07094776
Title: Evaluation of MG53 (TRIM72) Levels in Women With Polycystic Ovary Syndrome: An Observational Study
Acronym: PCOSMG53
Status: Enrolling by invitation | Type: Observational
Sponsor: Havva Betül Bacak (Other Government)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, M.D, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Other Study IDs: MG53GOP
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Insulin Resistance Syndrome
Keywords: MG53; TRIM72; Polycystic Ovary Syndrome; PCOS; Insulin Resistance; Metabolic Markers; ELISA; Cross-Sectional Study; HOMA-IR; SHBG; Androgen Index; Lipid Profile
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome; Insulin Resistance | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS Group: Women aged 18-45 years diagnosed with polycystic ovary syndrome (PCOS) based on Rotterdam criteria. A single blood sample is collected for MG53 and routine metabolic markers. No intervention is applied.
  Interventions: Other: No intervention (observational study)
- Healthy Controls: Women aged 18-45 years without PCOS or other chronic conditions. A single blood sample is collected for MG53 and routine metabolic markers. No intervention is applied.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study. No drugs, devices, or treatments are administered. Participants only provide a single blood sample for MG53 and routine metabolic measurements.

SUMMARY:
Purpose of the Study:

This study is being conducted to examine a protein called MG53 (also known as TRIM72) in women with polycystic ovary syndrome (PCOS). MG53 is involved in cell membrane repair and may play a role in insulin resistance, which is common in PCOS.

Study Procedures:

Women between 18 and 45 years of age will be invited to participate. The study population will include both women diagnosed with PCOS and healthy controls. A single blood sample (approximately 5 mL) will be collected from each participant. MG53 levels will be measured using an ELISA laboratory assay.

Significance of the Study:

Analysis of MG53 levels in relation to hormonal and metabolic markers may help determine whether MG53 is associated with insulin resistance and other characteristics of PCOS.

DETAILED DESCRIPTION:
Background:

Polycystic ovary syndrome (PCOS) is a common endocrine disorder in women of reproductive age and is often associated with insulin resistance and metabolic disturbances. MG53 (TRIM72) is a membrane repair protein that has been shown in some experimental studies to affect insulin signaling and glucose metabolism.

Rationale:

Because insulin resistance is a key feature of PCOS, investigating MG53 levels in women with PCOS may provide new insights into the pathophysiology of the syndrome. Understanding whether MG53 is elevated and how it correlates with metabolic and hormonal parameters could lead to new diagnostic or therapeutic approaches in the future.

Study Design:

This is an observational, cross-sectional, single-center study. A total of 128 participants will be included: 64 women diagnosed with PCOS (based on the Rotterdam criteria) and 64 healthy women as controls.

Procedures:

Each participant will undergo a single blood draw (approximately 5 mL). MG53 levels will be measured using an ELISA method. Routine laboratory markers associated with PCOS (including HOMA-IR, BMI, LH/FSH ratio, total testosterone, DHEA-S, SHBG, free androgen index, triglycerides, HDL, LDL, and total cholesterol) will also be recorded from standard clinical evaluations.

Data Analysis:

Statistical analysis will include normality testing (Kolmogorov-Smirnov), comparison of groups (Student's t-test or Mann-Whitney U test), and correlation analyses (Pearson or Spearman). Sample size was calculated using G*Power software.

Outcome Measures:

The primary outcome is the serum level of MG53. Secondary outcomes include the correlation between MG53 levels and metabolic/hormonal parameters.

Significance:

This study does not involve any investigational drug or device and poses minimal risk to participants. The findings may contribute to the understanding of metabolic pathways involved in PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 to 45 years
* Diagnosed with polycystic ovary syndrome (PCOS) according to Rotterdam criteria or healthy controls without PCOS
* Able and willing to provide informed consent

Exclusion Criteria:

Currently pregnant

* Presence of chronic systemic disease
* Use of metformin or any hormonal treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of women aged 18 to 45 years. One group includes women diagnosed with polycystic ovary syndrome (PCOS) based on the Rotterdam criteria, and the other group includes healthy female controls without PCOS or other chronic conditions. All participants will provide informed consent before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Serum MG53 level | Baseline (single time point at enrollment)
  Serum MG53 levels measured by ELISA in women with PCOS and healthy controls. Time Frame: At the time of blood draw (single measurement at enrollment)

SECONDARY OUTCOMES:
Correlation between MG53 levels and insulin resistance (HOMA-IR) | At the time of blood draw (single measurement at enrollment)
  Association between MG53 levels and HOMA-IR index derived from fasting glucose and insulin.
Correlation between MG53 levels and BMI | At the time of blood draw (single measurement at enrollment)
  Association between MG53 levels and body mass index (BMI).
Correlation between MG53 levels and hormonal parameters | At the time of blood draw (single measurement at enrollment)
  Association between MG53 levels and LH/FSH ratio, total testosterone, DHEA-S, SHBG, and free androgen index.
Correlation between MG53 levels and lipid parameters | At the time of blood draw (single measurement at enrollment)
  Association between MG53 levels and triglycerides, HDL-cholesterol, LDL-cholesterol, and total cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Enes S Coşkun, M.D., Principal Investigator — University of Health Sciences, Gaziosmanpaşa Training and Research Hospital
Locations (1):
- University of Health Sciences, Gaziosmanpaşa Training and Research Hospital, Gaziosmanpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study does not include a plan for public data sharing, and participant consent for data sharing has not been obtained.